CLINICAL TRIAL: NCT03367494
Title: A New Optical Sweat Test Method Based on a Citric Acid-derived Multi-halide Sensor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Robert Vender, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00008612
Record Dates: First submitted 2017-11-22; First posted 2017-12-08 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with Cystic Fibrosis (Other): Diagnostic
  Interventions: Diagnostic Test: Measurement of Sweat Chloride and Sweat Bromide
- Healthy Volunteers (Other): Diagnostic
  Interventions: Diagnostic Test: Measurement of Sweat Chloride and Sweat Bromide

INTERVENTIONS:
Diagnostic Test: Measurement of Sweat Chloride and Sweat Bromide — Sweat Chloride comparisons between ion exchange chromatography and fluorescence citrate-based sensors

SUMMARY:
Cystic Fibrosis (CF) is a hereditary multi-system disease affecting approximately 30,000n children and adults in the USA. The diagnosis of CF requires biochemical confirmation (either abnormal sweat chloride measurement and/or identification of two CF disease causing mutations) plus clinical symptomatology. Measurements of sweat chloride remain cumbersome and although most common methodology to confirm CF diagnosis with limitations especially in young children less than 6 months of age and in areas that lack ability for the complex testing. The study objectives of this current research proposal include: A) To expand upon previously obtained pilot study data "Evaluation of a fluorescent-based chloride sensor as an optical sweat test to diagnose cystic fibrosis" B) To add the exploratory measurement of sweat Bromide as a first in human assessment observation, C) To Evaluate the development of smartphone based point-of-care technology for chloride and bromide sensor measurements, D) To further expand the class of citrate-based sensors with improved fluorescence and sensing properties for the design of new fluorescence-based analytical and diagnostic solutions based on the automated multi-halide detection system, and E) To develop point-of-care systems that can successfully integrate into clinical settings to improve current practices and facilitate early detection of disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older capable of providing written informed consent AND
* Patients with an established diagnosis of Cystic Fibrosis (CF) OR Healthy volunteers

Exclusion Criteria:

* Participants under medications or with disorders known to cause a positive error in the sweat test will be excluded in the study. Common causes of positive error in sweat test are mineralocorticoid hormone therapy, adrenal insufficiency, glycogen storage diseases, hypothyroidism, hypoparathyroidism, nephrogenic diabetes insipidus, G6PD deficiency or ectodermal dysplasia OR
* Any other skin or soft tissue disorders that could affect obtaining the necessary volumes of sweat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Sweat chloride measurements in sweat samples via ion exchange chromatography | anticipated 12 months
  Sweat specimen samples obtained via pilocarpine iontophoresis will be measured for sweat chloride. Measurements for chloride will be determined by ion exchange chromatography measured in millimolar (mM).
Sweat chloride measurements in sweat samples via fluorescence quenching | anticipated 12 months
  Sweat specimen samples obtained via pilocarpine iontophoresis will be measured for sweat chloride. Measurements for the chloride will be determined by fluorescence citrate-based sensors, measured in millimolar (mM).
Sweat bromide measurements in sweat samples via fluorescence quenching | anticipated 12 months
  Sweat specimen samples obtained via pilocarpine iontophoresis will be measured for sweat bromide. Measurements for bromide will be determined by fluorescence citrate-based sensors, measured in millimolar (mM).

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
No personally identifiable information will be communicated to investigators at PSU-University Park. Sweat samples will be identified solely by code which code will be linked to personally identifiable information known only to Dr. Vender and which code will be kept in a locked office at Hershey Medical Center (HMC) Biomedical Research Building C5860. This code will contain participant (both CF patients and healthy volunteers): name, HMC medical record #, age, gender, date of sample, date of birth and sweat chloride/bromide results. In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared. Personally identifiable health information access (such as diagnosis, name, HMC medical record#, age, gender, date of birth) is specifically for Cystic Fibrosis patients. Medical records and health information will NOT be accessed for healthy control volunteers, however name, age, gender, date of birth will be recorded.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Zhang C, Kim JP, Creer M, Yang J, Liu Z. A smartphone-based chloridometer for point-of-care diagnostics of cystic fibrosis. Biosens Bioelectron. 2017 Nov 15;97:164-168. doi: 10.1016/j.bios.2017.05.048. Epub 2017 May 27. PMID 28595077
- [Background] Kim JP, Xie Z, Creer M, Liu Z, Yang J. Citrate-based fluorescent materials for low-cost chloride sensing in the diagnosis of Cystic Fibrosis. Chem Sci. 2017 Jan 1;8(1):550-558. doi: 10.1039/C6SC02962K. Epub 2016 Aug 30. PMID 28348728